CLINICAL TRIAL: NCT03577431
Title: A Phase I/II Drug Withdrawal Study of Alloantigen-Specific Tregs in Liver Transplantation (ITN073ST)
Brief Title: Liver Transplantation With Tregs at MGH
Acronym: LITTMUS-MGH
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN073ST
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Liver Transplant
Keywords: alloantigen-reactive Tregs ( arTreg); immunosuppression; operational tolerance
MeSH Terms: interventions — Leukapheresis; Blood Component Removal; Cyclophosphamide; Mesna; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- arTreg-CSB (Experimental): arTreg CSB: alloantigen-reactive T regulatory cells costimulatory blockade per protocol.
  The investigational product is donor alloantigen-specific T regulatory cells (arTreg-CSB). Supportive regimen for receipt of arTregs-CSB includes everolimus, leukapheresis, cyclophosphamide, and mesna.
  Participants will receive a single dose of Treg product (arTreg-CSB). The target dose is 2.5 to 125 x 10^6 total cells. arTreg-CSB will be administered as a single peripheral intravenous (IV) infusion over approximately 15 to 30 minutes.
  Note: Participants who receive at least the minimum Treg product (arTreg-CSB) dose of 1 to < 2.5 x 10^6 cells will be included in intent-to-treat analysis.
  Interventions: Biological: arTreg-CSB; Procedure: leukapheresis; Drug: cyclophosphamide; Drug: mesna; Drug: everolimus

INTERVENTIONS:
Biological: arTreg-CSB — Participants will receive a single dose of Treg product (arTreg-CSB). The target dose is 2.5 to 125 x 10^6 total cells. If a minimum arTreg-CSB dose of 1 to < 2.5 x 10^6 cells, the product will be infused. If the dose obtained after product manufacture is < 1 x 10^6 cells, the product will not be infused. When the dose obtained after product manufacture is > 125 x 10^6 cells, a dose aliquot will be prepared so that the administered dose will be ≤ 125 x 10^6 cells, and ≥ 2.5 to 125 x 10^6 total cells.
  Method of receipt: peripheral intravenous (IV) infusion, administered over 15 to 30 minutes.
  Other Names: donor alloantigen specific regulatory T cells; CD4+CD25+CD127[lo] Treg cells
Procedure: leukapheresis — Leukapheresis will be the method employed to recover peripheral blood mononuclear cells (PBMCs) from the allograft recipient. The recipient will undergo the procedure prior to initiating the cyclophosphamide conditioning regimen.
  Procedure 72 to 120 hours prior to Treg product (arTreg-CSB) IV infusion.
  Other Names: apheresis
Drug: cyclophosphamide — 40 mg/kg administered intravenously (IV) within 24 to 72 hours prior to Treg product (arTreg-CSB) infusion.
  Other Names: Cytoxan®
Drug: mesna — Mesna is administered intravenously to inhibit hemorrhagic cystitis induced by cyclophosphamide. Administration of mesna is per institutional practice with cyclophosphamide.
  Other Names: Mesnex®
Drug: everolimus — EVR, an immunosuppressant (IS), is approved by the FDA for the prophylaxis of allograft rejection in adults receiving a liver transplant. Between day 30 and wk. 48 post-transplant, participant evaluation for eligibility to be converted to an EVR-based IS regimen will occur.
  At the start of conversion from tacrolimus (TAC) to EVR IS:EVR will be started at 1.5 mg taken by mouth BID, with dose adjusted to achieve a trough blood level of 5-8 ng/mL. Once an EVR trough level of ≥ 5 ng/mL is achieved, baseline TAC dose will be reduced to achieve a trough level of 3-5 ng/mL.
  When target EVR and TAC levels are achieved/ maintained over two consecutive measurements, and liver function tests, ALT and GGT, are ≤50 U/L, participants will be considered successfully converted to EVR-based IS regimen. EVR doses will be administered, monitored and adjusted over time, per protocol.
  Other Names: EVR; Afinitor®; Zortress®

SUMMARY:
This is a single-center, prospective, open-label, non-randomized clinical trial exploring cellular therapy to facilitate immunosuppression withdrawal in liver transplant recipients.

DETAILED DESCRIPTION:
The researchers in this study plan to enroll 9 participants who will receive at least the target Treg product (arTreg-CSB) dose of 2.5 x 10^6 cells. Participants who receive at least 1 x 10^6 cells but < 2.5 x 10^6 cells as a result of low cell yield will be included in intent-to-treat (ITT) analysis.

Participants who successfully withdraw from all immunosuppression will undergo a research biopsy at 52 weeks following drug discontinuation to determine whether they meet the primary efficacy outcome of operational tolerance. Participants determined to be operationally tolerant will be followed until 104 weeks following drug discontinuation and have a research biopsy at that time to confirm that they remain operationally tolerant. Participants who fail drug withdrawal after 52 weeks but before 104 weeks will be followed until week 104 or 12 weeks after resuming immunosuppression, whichever is longer. The research biopsy at week 104 will be optional for these participants.

Participants who do not successfully withdraw from all immunosuppression will complete 104 weeks of High Intensity Safety Follow-up after failing immunosuppression withdrawal.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

Eligibility:

Recipient:

* Individuals must meet all of the following criteria to be eligible for this study:

  1. Able to understand and provide informed consent
  2. End-stage liver disease and listed for a living or deceased-donor primary solitary liver transplant
  3. Agreement to use contraception
  4. Positive Epstein-Barr virus (EBV) antibody test and
  5. In the absence of contraindication, vaccinations must be up to date per the DAIT Guidance for Patients in Transplant Trials (Refer to the Manual of Procedures)

     Living Donor:
* Living donors must meet all of the following criteria to be eligible for this study:

  1. Able to understand and provide informed consent
  2. Meets site-specific clinical donor eligibility requirements
  3. Meets donor eligibility manufacturing requirements within 7 days prior to blood collection for manufacturing and
  4. Willingness to donate appropriate biologic samples.

Deceased Donor:

Deceased donors must meet the following criteria for their recipients to be eligible for this study:

1. Meets site-specific clinical donor eligibility requirements and 2. Meets donor eligibility manufacturing requirements.

Note:

* There are several stages to this study.
* Eligibility is evaluated at many time points during the study to assess whether a participant is safe to proceed to the next study stage.

Exclusion Criteria:

Recipient:

* Individuals who meet any of the following criteria will not be eligible for this study:

  1. History of previous organ, tissue or cell transplant requiring or potentially requiring immunosuppression
  2. For cytomegalovirus (CMV) antibody negative recipients, a (CMV) antibody positive donor
  3. Known contraindication to cyclophosphamide or Mesna administration
  4. Serologic evidence of human immunodeficiency virus (HIV)-1/2 infection
  5. The need for chronic anti-coagulation that cannot be safely discontinued for a minimum of 1 week to safely perform a liver biopsy
  6. End stage liver disease secondary to autoimmune etiology (autoimmune hepatitis, primary biliary cirrhosis, or primary sclerosing cholangitis) or other contraindications to drug withdrawal
  7. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
  8. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the investigator, may interfere with study compliance
  9. Past or current medical problems, treatments or findings that are not listed above, which, in the opinion of the investigator, may:

     -- pose additional risks from participation in the study,
     * interfere with the candidate's ability to comply with study requirements, or
     * impact the quality or interpretation of the data obtained from the study.
  10. History of malignancy with a risk of recurrence judged by the investigator to be >1%, except for:

      -- hepatocellular carcinoma,

      -- completely treated in-situ cervical carcinoma, or

      -- completely treated basal cell carcinoma.
  11. Chronic use of systemic glucocorticoids or other immunosuppressives, or biologic immunomodulators.

      Living Donor:

      Living donors who meet the following criteria will not be eligible for this study:

  <!-- -->

  1. Any condition that, in the opinion of the investigator, may pose additional risks from participation in the study, may: -- interfere with the participant's ability to comply with study requirements or --impact the quality or interpretation of the data obtained from the study.

Deceased Donor:

Recipients of livers from deceased donors who meet the following criteria are ineligible for this study:

1. Any condition that, in the opinion of the investigator, may pose additional risks or may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) Attributed to the Investigational Product, arTreg-CSB | From arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  The number of AEs attributed to the investigational product, arTreg-CSB.
  AEs will be attributed to arTreg-CSB when the AE is reported with possible or related attribution to arTreg-CSB.
Severity of Adverse Events (AEs) Attributed to the Investigational Product, arTreg-CSB | From arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs attributed to the investigational product, arTreg-CSB.
  AEs will be attributed to arTreg-CSB when the AE is reported with possible or related attribution to arTreg-CSB.
  Grading according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Adverse Events (AEs) Attributed to the Investigational Product's Supportive Regimen (Leukapheresis, Cyclophosphamide and Mesna) | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  The number of AEs attributed to the investigational product's supportive regimen (leukapheresis, cyclophosphamide, and mesna).
  AEs will be attributed to the supportive regimen when the AE is reported with possible or related attribution to leukapheresis, cyclophosphamide, or mesna.
Severity of Adverse Events (AEs) Attributed to the Investigational Product's Supportive Regimen (Leukapheresis, Cyclophosphamide and Mesna) | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs attributed to the investigational product's supportive regimen (e.g., leukapheresis, cyclophosphamide, and mesna).
  AEs will be attributed to the supportive regimen when the AE is reported with possible or related attribution to leukapheresis, cyclophosphamide, or mesna.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Operationally Tolerant Participants | 52 weeks (±4 weeks) after the last dose of immunosuppression
  Operational tolerance is defined as:
  * Discontinuation of immunosuppression for 52 weeks,
  * Alanine aminotransferase (ALT) ≤ 50 U/L, and
  * A liver biopsy at 52 weeks (±4 weeks) after the last dose of immunosuppression that meets the criteria noted per protocol.
    * Liver histology will be assessed by central pathology.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) Attributed to Leukapheresis | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Number of AEs with possible or related attribution to leukapheresis.
Severity of Adverse Events (AEs) Attributed to Leukapheresis | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs with possible or related attribution to leukapheresis.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Adverse Events (AEs) Attributed to Cyclophosphamide | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Number of AEs with possible or related attribution to cyclophosphamide.
Severity of Adverse Events (AEs) Attributed to Cyclophosphamide | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs with possible or related attribution to cyclophosphamide.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Adverse Events (AEs) Attributed to Mesna | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Number of AEs with possible or related attribution to mesna.
Severity of Adverse Events (AEs) Attributed to Mesna | From ≤3 days prior to arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs with possible or related attribution to mesna.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Participants Who Experience ≥Grade 3 Infections Following arTreg-CSB Infusion | From arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Number of participants that experience ≥grade 3 infectious AEs status post arTreg-CSB infusion.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Biopsy-Proven Acute or Chronic Rejections | From arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Number of participants with biopsy-proven AR or CR. The diagnosis of biopsy-proven acute and chronic allograft rejection will be diagnosed in accordance with Banff global assessment criteria.
Severity of Biopsy-Proven Acute Rejections | From arTreg-CSB infusion through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of biopsy-proven AR at any time status post participant's receipt of arTreg-CSB infusion.
  Intensity of AR will be graded in accordance with the Banff global assessment criteria.
  Reference: Banff schema for grading liver allograft rejection: an international consensus document. Hepatology 1997;25:658-63.
Proportion of Participants with a Composite Outcome Measure of CR, Steroid Refractory AR, Retransplantation or Death Following Everolimus Conversion | From ≥30 days post-transplant through completion of study participation (Up to 4.5 years)
  The proportion of participants who develop ≥1 of the following events following initiation of everolimus conversion: refractory Acute Rejection (AR), Chronic Rejection (CR), undergo retransplantation, or die during study participation.
  Everolimus is FDA approved for use in liver and kidney transplantation for prophylaxis of organ rejection.
Number of AEs Attributed to Immunosuppression Withdrawal | From ≥30 days post-transplant through completion of study participation (Up to 4.5 years)
  Number of AEs possibly or definitely related to immunosuppression withdrawal.
Severity of AEs Attributed to Immunosuppression Withdrawal | From ≥30 days post-transplant through completion of study participation (Up to 4.5 years)
  Assessment of the intensity of AEs possibly or definitely related to immunosuppression withdrawal.
  Assessment of the intensity of AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events [NCI-CTCAE version 4.03].
Number of Participants who Develop a Malignancy | Day of transplant through completion of study participation (Up to 4.5 years)
  The number of participants that are diagnosed with malignancy, any type.
Number of Participants who Develop de novo Donor Specific Antibodies (DSA) | Baseline (pre liver transplant) through completion of study participation (Up to 4.5 years)
  A de novo donor-specific alloantibody (DSA) is a newly developed alloantibody that targets the donor organ. Alloantibodies are important mediators of acute and chronic rejection.
  This measure is calculated as time from transplant until the earliest time of development of any de novo DSA.
Number of Participants who Develop de novo non-DSA HLA Antibodies | Baseline (pre liver transplant) through Completion of Study Participation (Up to 4.5 years)
  The number of participants who, following liver transplant, develop anti-donor HLA alloantibodies defined by the presence of anti-HLA IgG antibodies.
Proportion of Participants who, Though Clinically Stable for 52 Weeks after Discontinued Immunosuppression per Protocol Schedule, do not Fulfill the Study Definition of Tolerance | Post-Transplant through Completion of Study Participation (Up to 4.5 years)
  Proportion of participants who have discontinued immunosuppression for 52 weeks, but have:
  * either an ALT greater than 50 U/L or
  * a liver biopsy at 52 weeks that does not show rejection but does not meet the biopsy criteria for operational tolerance (Reference: Demetris AJ, Bellamy C, Hubscher SG, et al. 2016 Comprehensive Update of the Banff Working Group on Liver Allograft Pathology: Introduction of Antibody-Mediated Rejection. Am J Transplant 2016).
Duration of Operational Tolerance | Post-transplant through Completion of Study Participation (Up to 4.5 years)
  Defined as the time from achievement of the primary endpoint to immunosuppression reinitiation or to the end of trial participation.
  Inclusion in this analysis is limited to those participants classified as operationally tolerant for the primary outcome measure.
Proportion of Participants who Successfully Discontinue Tacrolimus | Post-transplant through Completion of Study Participation (Up to 4.5 years)
  Proportion of participants who, per protocol:
  * fulfill eligibility for tacrolimus withdrawal,
  * subsequently achieve their last dose of tacrolimus,
  * remain tacrolimus-free for ≥12 weeks,
  * their liver function test, ALT is ≤50 U/L,
  * and their liver biopsy performed between 12 to 26 weeks status post the last dose of tacrolimus fulfills biopsy findings* for minimization of immunosuppression.
    * Biopsy findings: Liver histology will be assessed by central pathology. Biopsy findings for minimization of immunosuppression, per protocol. Reference: Demetris AJ, Bellamy C, Hubscher SG, et al. 2016 Comprehensive Update of the Banff Working Group on Liver Allograft Pathology: Introduction of Antibody-Mediated Rejection. Am J Transplant 2016.

CONTACTS AND LOCATIONS:
Overall Officials: James F. Markmann, MD, PhD, Study Chair — University of Pennsylvania Medical Center: Transplantation
Locations (1):
- Massachusetts General Hospital: Transplantation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network web site — http://www.immunetolerance.org